CLINICAL TRIAL: NCT02700568
Title: Evaluation of the Safety and Efficacy of Axitinib in Metastatic Renal Cell Carcinoma Patients With Favorable Prognostic Factors
Brief Title: Axitinib in Metastatic Renal Cell Carcinoma Patients With Favorable Prognostic Factors
Acronym: FavorAx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAVORAX-1
Record Dates: First submitted 2016-01-18; First posted 2016-03-07 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Carcinoma, Renal Cell; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- axitinib (Experimental): Patients will receive axitinib.
  Interventions: Drug: axitinib

INTERVENTIONS:
Drug: axitinib — Initial dose of axitinib: 5 mg orally twice a day. Maintenance dose of axitinib: Increase or decrease dose based on individual safety and tolerability. Dose range of axitinib: 2 to 10 mg twice a day.
  Other Names: Inlyta

SUMMARY:
Aim of the FavorAx study is to evaluate preliminary efficacy and safety of Axitinib in metastatic renal cell carcinoma patients with favorable IMDC prognostic factors who had progressed on sunitinib or pazopanib in the first-line setting.

DETAILED DESCRIPTION:
Axitinib is a tyrosine kinase inhibitor of vascular endothelial growth factor receptor, platelet-derived growth factor receptor-α, and c-kit. The trial of comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS) was an international randomized Phase III study designed for registration purposes. This trial randomized 723 metastatic renal cell carcinoma patients with any prognostic features to axitinib or sorafenib in the second-line setting and demonstrated significant clinical benefit of axitinib.

Aim of present FavorAx study is to evaluate preliminary efficacy and safety of Axitinib in metastatic renal cell carcinoma patients with favorable IMDC prognostic factors who had progressed on sunitinib or pazopanib in the first-line setting.

ELIGIBILITY:
Principle Inclusion Criteria:

* Histologic confirmation of Renal cell carcinoma with a clear cell component
* Patients must have measurable disease
* Previous treatment with sunitinib or pazopanib
* Favorable prognosis according to IMDC criteria
* Must have available tumor tissue for submission
* Subjects must also meet various laboratory parameters for inclusion
* Patients must give written informed consent prior to initiation of therapy

Exclusion Criteria:

* Any underlying medical condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events
* Patients who have history of uncompensated diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 10 months

SECONDARY OUTCOMES:
Objective response rate | 24 months
Overall survival | 24 months
Rate of treatment-related serious adverse events | 24 months
  Number of participants with treatment-related serious adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Tsimafeyeu, MD, Study Director — Kidney Cancer Research Bureau
Locations (15):
- Russia (15):
  - Demchenkova Marina Viktorovna, Irkutsk
  - Semenov Andrey Vladimirovich, Ivanovo
  - Mikhailova Nadezhda Vasilievna, Kazan'
  - Eskerov Kurban Abdulmutalibovich, Kirov
  - Zukov Ruslan Aleksandrovich, Krasnoyarsk
  - Ovchinnikova Elena Georgievna, Nizhny Novgorod
  - Guseva Irina Vasilievna, Penza
  - Vladimirova Lyubov Yur'evna, Rostov-on-Don
  - Zolotoreva Tatiana Gennadievna, Samara
  - Katkov Alexey Aleksandrovich, Saratov
  - Ivannikov Andrey Andreyevich, Tambov
  - Usynin Evgeny Anatolievich, Tomsk
  - Evstegneyeva Irina Vladimirovna, Tver'
  - Khmelevsky Andrey Anatolievich, Ufa
  - Gurina Ludmila Ivanovna, Vladivostok

IPD SHARING:
Plan to Share IPD: Undecided